CLINICAL TRIAL: NCT00810030
Title: Select A Multi-centre Randomised Prospective Open-label Study to Investigate the Efficacy & Safety of a Standardised Correction Dosage Regimen of i.v. Ferric Carboxymaltose Versus Iron Sucrose for Treatment of Iron Deficiency Anaemia in Patients With Inflammatory Bowel Disease
Brief Title: FERINJECT for Correction of Anaemia in IBD Patients, FER-IBD-COR
Acronym: FER-IBD-COR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: Parexel (Industry); ClinStar, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-IBD-07-COR
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Inflammatory Bowel Disease; Anemia; Iron Deficiency; Iron-Deficiency Anemia; Crohn's Disease; Ulcerative Colitis
Keywords: ferric carboxymaltose; iron sucrose; Iron-Deficiency Anemia; Crohn's Disease; Ulcerative Colitis; Ferritin; Transferrin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anemia; Iron Deficiencies; Anemia, Iron-Deficiency; Crohn Disease; Colitis, Ulcerative | interventions — ferric carboxymaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FERINJECT® (Ferric carboxymaltose) (Experimental)
  Interventions: Drug: Ferric carboxymaltose
- VENOFER® (Iron Sucrose) (Active Comparator)
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Dosage form: 5% w/v iron containing 50 mg iron per mL, as sterile solution of FERINJECT® in water for injection. In case of drip infusion FERINJECT® (10 to 20 ml) must be diluted only in sterile 0.9% sodium chloride (max 250 ml) FERINJECT® will be administered via i.v. drip infusion. Minimum administration time 15 minutes Dosage: 500 mg, 1000 mg, 1500 mg, according to patients' Hb and body weight
  Other Names: FERINJECT®
  Arms: FERINJECT® (Ferric carboxymaltose)
Drug: Iron Sucrose — VENOFER® will be administered via i.v. drip infusion, diluted only in sterile 0.9% sodium chloride solution as follows:
  • 10 mL Venofer® (200 mg iron) in maximum 200 mL sterile 0.9% sodium chloride solution in at least 30 minutes.
  The first 25 mL of solution should be infused as a test dose over a period of 15 minutes. If no adverse reactions occur, use infusion rate no more than 50 mL in 15 minutes.
  The individual iron deficit will be calculated using the modified formula of Ganzoni.
  If the patient's body mass index is >25, a normalised weight will be used for the calculation of iron deficit. Normalised weight = 25 x height [m] x height [m].
  The calculated cumulative VENOFER® dose is to be rounded up or down to the nearest 200 mg.
  Patients will receive one 200 mg VENOFER® infusion, twice a week, up to 11 times (max dosage 2200 mg), depending on their calculated iron deficit.
  Other Names: VENOFER®
  Arms: VENOFER® (Iron Sucrose)

SUMMARY:
The purpose of this study is to determine how safe, tolerable and effective the new standardised dosage regimen of FERINJECT® infusions is, compared with a well established intravenous iron treatment.

DETAILED DESCRIPTION:
Anaemia in inflammatory bowel disease is mainly attributed to iron deficiency. The main cause of anaemia in IBD patients is chronic blood loss. This means that the iron storage depot in IBD patients is always low and should be replenished. Oral iron therapy is the first choice in many cases because of its safety and economy. However, in patients with gastrointestinal bleeding, the effectiveness of oral therapy is reduced. Additionally, oral iron preparations are frequently associated with gastrointestinal adverse reactions.

According to European Guidelines, the preferred route of iron supplementation in IBD is intravenous. Absolute indications for intravenous iron include severe anaemia (Hb <10 g/dL). The current study is a part of a programme investigating the efficacy and safety of FERINJECT®, a new formulation of parenteral iron (5% weight per volume iron containing ferric carboxymaltose in a solution of water for injection).

The efficacy and safety of FERINJECT® were investigated in a prospective, randomised, controlled study conducted in IBD patients. According to the results of this study, FERINJECT® provides a faster Hb response, a higher increase in iron storage and a better patient tolerance compared to oral preparations. In this study, the iron amount required was calculated according to the Ganzoni formula, where 500 mg is the amount of storage iron. To simplify the treatment and to make the treatment more effective, a new standardised dosage regimen was created. The current study is designed to assess whether this new standardised dosage regimen of i.v. FERINJECT® is as safe and effective as the currently used individually calculated dosage regimen.

The efficacy and safety of the new standardised dosage regimen of FERINJECT® will be compared with an already established, well-known treatment of IDA with iron sucrose (VENOFER®). Iron sucrose (VENOFER®) is assessed to be effective and well-tolerated in the treatment of IDA in IBD patients.

The study is a phase IIIb, multi-centre, randomised, prospective, open-label, controlled study performed at 83 study centres in 14 European countries.

The primary objective of the study is to evaluate the non-inferiority in efficacy of a standardised dosage regimen of FERINJECT® compared to individually calculated dosage regimens of VENOFER® in the correction of IDA in patients with IBD in remission. The secondary objective is to evaluate the safety and tolerability of a standardised correction dose regimen of FERINJECT®.

Approximately 420 patients will be randomised (1:1 randomisation) to receive treatment with either a standardised correction dosage regimen of FERINJECT® or individually calculated dosage regimens of VENOFER®.

Screening will start between 14 and 7 days before the first infusion is administered. Baseline assessments will be performed on Day 1 before the first infusion.

During the screening period, patients will be selected based on eligibility criteria. Patients who meet all of the inclusion criteria and none of the exclusion criteria will undergo baseline assessments at Baseline (Day 1) prior to the first dose of study medication.

Patients randomised to the FERINJECT® group will receive between 500 mg and 2000 mg of FERINJECT®, according to their Hb and body weight, in up to 3 infusions. The maximum infused weekly dose of will be 1000 mg. For patients in the VENOFER® group, the individual iron deficit will be calculated per individual using the modified formula of Ganzoni. Patients will receive one infusion of 200 mg of VENOFER® twice a week, up to 11 infusions, depending on their calculated iron deficit. Due to the relatively large doses of iron being administered, patients will be monitored carefully throughout the study for symptoms of iron overload.

All patients will return for assessment of efficacy and safety at Weeks 4, 8, and 12. The maximum study duration for a patient is 14 weeks. Patients who are not anaemic at Week 12 will be invited to continue to participate in a maintenance study (FER-IBD-07-MAIN), i.e. a study of FERINJECT® versus placebo to determine if the treatment of iron deficiency can prevent the recurrence of anaemia.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent.
* Patients ≥18 years of age suffering from mild IBD (CD/UC) or in remission (mild IBD defined as CDAI score <220, or CAI score ≤7, remission defined as CDAI score <150, or CAI score ≤4).
* Hb 7-12 g/dL (female) or 7-13 g/dL (male).
* Ferritin <100 μg/L.
* Normal levels of vitamin B12 and folic acid.
* Females of child-bearing potential must have a negative urine pregnancy test at screening and be practising an acceptable method of birth control during the study and for up to 1 month after the last dose of study medication.

Exclusion Criteria

* Chronic alcohol abuse (alcohol consumption >20 g/day).
* Presence of portal hypertension with oesophageal varices.
* History of erythropoietin, intravenous or oral iron therapy, or blood transfusion in 4 weeks prior to screening.
* Known hypersensitivity to FERINJECT®.
* History of acquired iron overload.
* Myelodysplastic syndrome.
* Pregnancy or lactation.
* Known active infection, clinically significant overt bleeding, active malignancy.
* Known chronic renal failure. Vifor Pharma - Vifor (International) Inc Clinical Study Protocol inc. Amendments 1 and 2 Protocol Number: 93842, FER-IBD-07-COR CONFIDENTIAL Final 20 of 48 10 December 2008
* Surgery with relevant blood loss (defined as Hb drop <2 g/dL) in the last 3 months prior to screening or planned surgery within the following 3 months.
* Chronic liver disease or increase of liver enzymes (alanine aminotransferase ([ALT], aspartate aminotransferase [AST]) >3 times the upper limit of normal range.
* Known human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Inability to fully comprehend and/or perform study procedures in the investigator's opinion.
* Participation in any other interventional study within 1 month prior to screening.
* Body weight <35 kg.
* Significant cardiovascular disease, including myocardial infarction within 12 months prior to study inclusion, congestive heart failure NYHA (New York Heart Association) grade III or IV, or poorly controlled hypertension according to the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of responders with respect to the baseline Hb value. | 12 weeks post baseline
  Number of responders (Hb increase ≥2 g/dL) with respect to the baseline Hb value.

SECONDARY OUTCOMES:
Number of patients whose Hb increased ≥2 g/dL or who reached normal Hb levels at Week 12. | 12 weeks post baseline
  The number of patients who achieved increase of Hb ≥2 g/dL or the normal range of Hb value of Hb ≥12 (female) or ≥13 (male) g/dL) at Week 12.
Change in disease activity (CDAI, CAI, C-reactive protein [CRP]). | 12 weeks post baseline
  Change in disease activity (Crohn's Disease Activity Index [CDAI], Colitis Activity Index [CAI], C-reactive protein [CRP]) at Week 12.
The number of patients at Week 12: TfS: 20 to 50%. | 12 weeks post baseline
  The number of patients at Week 12: TfS: 20 to 50%.
The number of non-anaemic patients at Week 12 | Week 12 post baseline
  The number of non-anaemic patients at Week 12: Hb ≥12 (female) or ≥13 (male) g/dL.
The number of patients with ferritin >100 µg/L at Week 12. | 12 weeks post baseline
  The number of patients with ferritin >100 µg/L at Week 12.
Maximum increase in Hb, serum ferritin and TfS. | 12 weeks post baseline
  Maximum increase in Hb, serum ferritin and TfS.
The number of patients at achieving Hb ≥12 (female) or ≥13 (male) g/dL and ferritin >100 µg/L at Week 12. | 12 weeks post baseline
  The number of patients at Week 12: Hb ≥12 (female) or ≥13 (male) g/dL and ferritin >100 µg/L.
The number of patients withdrawal from study due to protocol procedure. | 12 weeks post baseline
  The number of patients withdrawal from study due to protocol procedure.
The number of responders (Hb increase ≥2 g/dL) with respect to treatment of underlying disease. | 12 weeks post baseline
  The number of responders (Hb increase ≥2 g/dL) with respect to treatment of underlying disease.
The number of patients with Hb baseline value ≤10 g/dL who achieved Hb increase ≥2 g/dL and the number of patients with Hb baseline value >10 g/dL who achieved Hb increase ≥2 g/dL. | 12 weeks post baseline
  The number of patients with Hb baseline value ≤10 g/dL who achieved Hb increase ≥2 g/dL and the number of patients with Hb baseline value >10 g/dL who achieved Hb increase ≥2 g/dL.
Change in health-related quality of life (QoL) from baseline to Week 12 using the Short Form (SF)-36, version 2 and IBDQ. | 12 weeks post baseline
  Change in health-related quality of life (QoL) from baseline to Week 12 using the Short Form (SF)-36, version 2 and IBDQ.
The number of patients out of work due to anaemia or IBD. | 12 weeks post baseline
  The number of patients out of work due to anaemia or IBD.
Days out of hospital. | 12 weeks post baseline
  Days out of hospital.
Hospitalisation rate | 12 weeks post baseline
  Hospitalisation rate (hospitalisation due to anaemia and/or IBD).
Adverse events: type, nature, incidence and outcome. | 12 weeks post baseline
  Adverse events: type, nature, incidence and outcome.
Vital signs (blood pressure, pulse rate and bw). | 12 weeks post baseline
  Vital signs (blood pressure, pulse rate and bw).
Electrocardiogram. | 12 weeks post baseline
  Electrocardiogram.
Change in laboratory parameters (haematology, clinical chemistry, iron status, urinalysis). | 12 weeks post baseline
  Change in laboratory parameters (haematology, clinical chemistry, iron status, urinalysis).
Physical examination. | 12 weeks post baseline
  Physical examination.
The number of responders (Hb increase ≥2 g/dL) with respect to the baseline Hb value. | 12 weeks post baseline
  The number of responders (Hb increase ≥2 g/dL) with respect to the baseline Hb value.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gasche, Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- AKH Vienna, University clinic of Int Medizin III, Vienna, Austria